CLINICAL TRIAL: NCT05138172
Title: Forced Air Heating to Prevent Hypothermia During Endoscopic Retrograde Cholangiography
Acronym: FAIRHEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: FAIRHEC
Record Dates: First submitted 2021-11-08; First posted 2021-11-30 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Temperature Management During Sedation for Endoscopic Retrograde Cholangiography
Keywords: sedation; endoscopic retrograde cholangiography; temperature managment; hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedation without forced air heating temperature management (Placebo Comparator): Sedation without forced air heating temperature management = present standard in sedation during endoscopic retrograde cholangiography (ERC)
  Interventions: Device: Forced Air Heating Temperature control "Twinwarm II"
- Sedation with forced air heating temperature management (Experimental): Sedation without forced air heating temperature management = proposed new standard in sedation during endoscopic retrograde cholangiography (ERC)
  Interventions: Device: Forced Air Heating Temperature control "Twinwarm II"

INTERVENTIONS:
Device: Forced Air Heating Temperature control "Twinwarm II" — For this purpose, we will use a device that is already routinely used in all operation rommss at MHH, the so-called "warm air device Twinwarm, Generation III". This device has a valid CE mark and will be used according to its purpose "pre-, intra- and postoperative maintenance of the normothermic body temperature of the patient". The device will be used strictly according to the existing in-house SOP "Heat Management" of 04/2021 of the Department of Anesthesiology and Intensive Care Medicine of the MHH.
  Convective air heating has been shown to be effective in many studies and can be used flexibly with a variety of different ceiling models.

SUMMARY:
The aim of this prospective observational study is to evaluate the role of a convective warming blanket to prevent hypothermia during sedation for an endoscopic retrograde cholangiography (ERC).

DETAILED DESCRIPTION:
During endoscopic retrograde cholangiography (ERC), deep medical sedation of the patient is routinely perform. Since ERC is a complex examination and in addition sometimes several intervention steps are necessary (bougienage, dilatation, brush cytology, specimen collection, insertion of plastic and metal stent prostheses), the sedation time is almost always > 30min, in many cases even up to one hour or longer. These patients are at risk for developing hypothermia (drop in core body temperature below 36 degrees Celsius).

It is well known from anesthesiologic research that even moderate perioperative hypothermia, however, can have potentially serious complications. These include increased mortality, cardiac complications such as arrhythmias and infarctions, coagulation disorders, and increased transfusion requirements and wound infections. Changes in serum concentrations of potassium and peripheral vasoconstriction with decrease in subcutaneous partial pressure of oxygen are also clinically important side effects of perioperative hypothermia.

However, the current 2014 German S3 guideline "Sedation in gastrointestinal endoscopy" does not mention peri- or intra-interventional temperature measurement or temperature management.

The aim of this prospective observational study is to evaluate the role of a convective warming blanket to prevent hypothermia during sedation for an ERC. From the description of various clinical endpoints, we seek to obtain sufficient evidence to support routine use of such a system in ERC examinations. This study has the potential to set the new standard for modern sedation during ERC interventions that recognizes the risk of hypothermia and identifies a strategy to avoid it.

For this purpose, we will use a device, that is already routinely used in all operation rooms in Germany, the so-called warm air device "Twinwarm, Generation III". This device has a valid CE mark and will be used according to its purpose "pre-, intra- and postoperative maintenance of the normothermic body temperature of the patient". The device will be used strictly in accordance with the existing in-house SOP "Heat Management" of 04/2021 of the Department of Anesthesiology and Intensive Care Medicine of Hannover Medical School (MHH).

ELIGIBILITY:
Inclusion criteria:

* Indication to receive repeat (≥ 2 expected interventions) endoscopic retrograde cholangiography (ERC) (The following underlying conditions may be considered as indications for repeat ERC to be performed:
* Primary sclerosing cholangitis (PSC)
* Ischemic type biliary lesion (ITBL) after liver transplantation (LTX)
* Anastomotic stenosis after LTX
* Secondary sclerosing cholangitis (SSC))
* necessary intravenous medical sedation is expected to be required >30min (female and male, age ≥ 18 years).

Exclusion Criteria:

* Patients < 18 years
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Highest absolute change of T from baseline at any time during intervention as well as at the end of intervention | During Intervention
  Primary Endpoint

SECONDARY OUTCOMES:
Percentage of patients with a reduction of T from baseline more than 1 degree Celsius at any time during intervention as well as at the end of intervention | During Intervention
  Key Secondary Endpoint
Percentage of patients with a reduction of T below 36 degree Celsius at any time during intervention as well as at the end of intervention | During Intervention
  Percentage of patients with a reduction of T below 36 degree Celsius
Hemodynamic stability | During Intervention
  Mean arterial pressure (MAP)
  * Lowest absolute MAP (mmHg)
  * Percentage of patients with a reduction of MAP of at least 25% from baseline
  * Absolute change of MAP below 65mmHg from baseline
  Heart Rate:
  * Relative difference: Percentage of patients with an increase of HR of at least 25% from baseline
  * Percentage of patients with a increase of heart rate > 100bpm
  Intravenous fluids:
  * Percentage of patients (%) needing intravenous fluid support for hemodynamic stability
  * Cumulative total Volume (ml) of intravenous fluid support
  Vasoactive substances:
  - Percentage of patients (%) needing vasoactive substance support
Respiratory Stability | During Intervention
  peripheral Oxygen Saturation (O2-Sat)
  - Percentage of patients with a reduction of O2-Sat below 90%
  Oxygen support:
  * Percentage of patients needing > 2l/min oxygen
  * Maximum needed flow (l/min) of oxygen delivery
  Further adverse events:
  * Percentage of patients (%) needing mask ventilation
  * Percentage of patients (%) with need for Guedel or Wendel tube insertion
Subjective Patient Satisfaction | 6 hours after intervention
  Subjective Freezing (VAS 0-10 points, with higher scores indicating more intense freezing)
  Quality of Recovery (QoR) Score by Myles et al. (Use of the German Modifikation by Eberhart et al) with score ranging from 0 to 18 points and higher scores indicating more discomfort with anesthesia
  modified DGAI Score with score ranging from 0 to 9 points and higher scores indicating more discomfort with anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared on reasonable request.